CLINICAL TRIAL: NCT05706584
Title: The Effect of Metaverse-Based Nursing Skills Laboratory on Teaching Pediatric Nursing Practice Skills
Brief Title: The Effect of Metaverse-Based Nursing Skills Laboratory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gulay Turk, PHD Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MedipolU-0001-Gturk
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Premature
Keywords: nursing; pediatric; metaverse; skill laboratory
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study was planned with a mixed method consisting of single-blind randomized controlled experiment and focus group interview methods. The research was planned to be carried out during the pediatric nursing course period between 2023-2024 Fall Semester October-December. Participants will be students taking a pediatric nursing course. Scales and Forms to be used in the Study; Informed Consent and Demographic Data Collection Form, Expert Opinion Form, Proficiency Scale for Nursing Students, Augmented Reality Applications Attitude Scale, Pre and Post Test, Student Case Form, Orogastric Catheter Application Procedure Steps Checklist and Distance Education Satisfaction Scale of university life.
Who Masked: Participant
Masking Description: With the simple randomization method, students will be assigned to the experimental and control groups. Even the last digit of the student number will be randomized to the experimental group and odd ones will be randomized to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control grup (skill lab.) (No Intervention): After the control group was determined from the students attending the child health and diseases nursing course in the 2023 -2024 fall semester.
  * The control group will be informed and approved.
  * The control group will be pre-tested
  * The control group will go to the skill laboratory.
- experimental group (metaverse skill lab.) (Experimental): After the experimental group was determined from the students attending the pediatric health and diseases nursing course in the fall semester of 2023-2024, respectively.
  * Pre-test will be applied to the experimental group.
  * Informed consent and demographic data collection form will be obtained from the experimental group.
  * The experimental group will be informed about the metaverse and approval will be obtained.
  * Premature infant nutrition training will be given to the experimental group in a metaverse-based skill laboratory environment.
  * The experimental group will enter the metaverse skill laboratory environment one by one, select their avatar and switch to the patient room in the environment,
  * The experimental group will evaluate the feeding pattern of the premature baby on the scenario given first in the metaverse-based skills laboratory.
  Interventions: Other: control grup (skills lab.) and experimental group (mateverse skill lab.)

INTERVENTIONS:
Other: control grup (skills lab.) and experimental group (mateverse skill lab.) — The universe of the study consists of students (N: 190) who took a pediatric nursing course in the 3rd year of the Teaching Department at Istanbul Medipol University. The sample of the study will consist of the students who took the 3rd year child health and diseases nursing course in the nursing department, accepted the study, and met the study criteria. It will try to reach the universe where the sample selection of the research will not be made. With the simple randomization method, students will be assigned to the experimental and control groups. Even the last digit of the student number will be randomized to the experimental group and odd ones will be randomized to the control group
  Arms: experimental group (metaverse skill lab.)

SUMMARY:
Depending on the education system, the increasing number of students, inadequate practice/skill laboratories, a small number of lecturers and students with limited time in the clinic have a negative impact on obtaining appropriate clinical experience. The virtual learning environment experience will prepare the student for the clinic in the most realistic way and will reduce the risk of errors in clinical care and treatment. In light of this information, presenting the learning environment of the future to the student will prepare the student both in the clinical practice area and in the professional environment as self-confident and highly equipped The study was planned with a mixed method consisting of single-blind randomized controlled experiment and focus group interview methods. The research was planned to be carried out during the pediatric nursing course period between 2023-2024 Fall Semester October-December. Participants will be students taking a pediatric nursing course. Scales and Forms to be used in the Study; Informed Consent and Demographic Data Collection Form, Expert Opinion Form, Proficiency Scale for Nursing Students, Augmented Reality Applications Attitude Scale, Pre and Post Test, Student Case Form, • Focus Group Interview Form and Distance Education Satisfaction Scale of university life.

The universe of the research consists of all students who take and continue the 2023 - 2024 fall term child health and diseases nursing course (N: 190). It will try to reach the universe where the sample selection of the research will not be made.

To measure the learning efficiency of pediatric nursing students in infant orogastric tube care application in two different skill laboratories, considering the feeding pattern from Gordon's Functional Health patterns. (University skills lab and metaverse-based clinical skills lab) As a result, the learning levels of the students in the metaverse-based clinical skills laboratory environment will be higher than in the skills laboratory. It will also increase the student's self-confidence in the field of pediatric nursing practice.

DETAILED DESCRIPTION:
Depending on the education system, the increasing number of students, inadequate practice/skill laboratories, a small number of lecturers, and students with limited time in the clinic have a negative impact on obtaining appropriate clinical experience. In addition, from the perspective of Bloom's taxonomy, learning; reminding, understanding, applying, analysing, evaluating and creating. Due to the limitations in clinical applications, students often cannot progress to advanced stages from the application part of Bloom's taxonomy.

Today, clinical application areas are limited within the structure of the health care system. In addition, considering the developments in technology, it is necessary to include innovative approaches in education in line with the expectations of students coming to higher education. Therefore, simulation-based learning has been one of the effective methods in preparing nursing students for the clinic and profession with knowledge and skills.

Use of virtual reality simulation among nursing students and working nurses: Among the three learning outcomes (skill-based, cognitive, and affective) in a systematic review, virtual worlds are most effective in improving cognitive outcomes such as theoretical knowledge. This situation suggests that virtual worlds can be used as an alternative or complementary method in teaching theoretical knowledge in nursing education and that a learning environment should be designed in accordance with the innovations brought by technology for clinical applications in nursing education. In addition, the prevalence and demand of online/distance education systems in the education system and the necessity of using them in extraordinary situations increase the necessity of a technological learning environment. Virtual reality, augmented reality, artificial intelligence and metaverse-based simulation environment are among the most suitable methods that can be chosen to develop learning, decision making, critical thinking and clinical skills.

Metaverse is Augmented Reality or Cross Reality (XR) based on technologies that enable multi-sensory interactions with virtual environments, digital objects, and people. XR includes Virtual Reality (VR), Augmented Reality (AR), and Mixed Reality (MR) (Milgram et all., 1994). The representative accuracy of the XR system is ensured by stereoscopic displays capable of transmitting depth perception. XR systems allow active interaction with virtual items through the use of motion controllers. These are handheld input devices with a handle, buttons, triggers, and thumbsticks. Using controllers, users can touch, hold, manipulate and operate virtual objects. This ability enables them to be active in any educational experience (such as nursing care).

The importance of this study is to provide an evidence-based virtual education environment to the literature and to ensure that it is ready for extraordinary situations in the field of education (such as distance education during the pandemic period). This should be done by designing and developing a virtual learning environment. While aiming to make this environment in the study, was based on evidence. The use of Gordon's Functional Health Patterns in the design of the virtual learning environment is important in terms of meeting the patient and starting the nursing process when the student first enters the clinical environment The virtual learning environment experience will prepare the student for the clinic in the most realistic way and will reduce the risk of errors in clinical care and treatment. In the light of this information, presenting the learning environment of the future to the students will prepare the student both in the clinical practice area and in the professional environment as self-confident and highly equipped.

The aim of the study is to analyze two different skill laboratory experiences of pediatric nursing students (the course and practice laboratory experiences they took during the formal education period and the lessons and practice experiences they received in the metaverse -based skill laboratory environment) within the feeding pattern of Gordon's Functional Health Patterns, through the example of orogastric tube application in the premature baby is to compare. The study was planned with a mixed method consisting of single-blind randomized controlled experiment and focus group interview methods.

Objectives of The Research

1. To design a metaverse-based clinical skills environment that will provide practical skills,
2. control and experimental groups in simulation environments (control group; skill laboratory, experimental group; metaverse -based clinical skills laboratory environment),
3. Taking the experimental group into a focus group interview,
4. Evaluating the success and satisfaction of the experimental / control groups

Questions of The Research

1. the clinical practice skills of the 3rd year child health and diseases nursing students be gained in the metaverse-based clinical skills laboratory environment?
2. Metaverse of 3rd-grade child health and diseases nursing students What will be the success rate when comparing student achievement in clinical practice courses and a clinical skills laboratory-based environment?
3. Can it be used as a teaching method in distance education for 3rd-grade child health and disease nursing students?

Hypotheses of the Study

1. H0: The education level of the 3rd-grade child health and diseases nursing students in the metaverse-based clinical skills laboratory environment is lower than the education level in the skill laboratory.
2. H1: The education level of the 3rd year pediatric nursing students in the metaverse-based clinical skills laboratory environment is higher than in the skill laboratory.

AIM To measure the learning efficiency of pediatric nursing students in infant orogastric tube care practice in two different skill laboratories, taking into account the feeding pattern from Gordon's Functional Health patterns. (University skills laboratory and metaverse-based clinical skills laboratory) The study was planned with a mixed method consisting of single-blind randomized controlled experiment and focus group interview methods.

Research time 2023-2024 Fall Semester is the period of pediatric nursing course between October and December. Participants are students taking pediatric nursing course.

Ethical Considerations and Limitations of Research The study will be initiated by obtaining informed consent from the students who took the pediatric nursing course during the academic year. Institutional and ethical committee permissions will be obtained. (No: E-31034136-302.08.01-649) The research was carried out within the framework of the Declaration of Helsinki, good clinical guide practices and the law on the protection of personal information will be followed.

The limitations encountered in this study are listed below.

* The sample of the research is limited to the students who take a pediatric nursing course in the Department of Nursing at the Faculty of Health Sciences of Medipol University.
* Expert opinions on the metaverse-based clinical skills laboratory will be obtained from academic staff who are experts in the field of pediatric nursing and engineering.
* Experience of participants in the designed metaverse-based clinical skills laboratory; It is limited to the features of the virtual reality glasses and equipment (headset, controller, etc.) used within the scope of the study.

Sample of the Study The universe of the study consists of students (N: 190) who took a pediatric nursing course in the 3rd year of the Teaching Department at Istanbul Medipol University. The sample of the study will consist of the students who took the 3rd year child health and diseases nursing course in the nursing department, accepted the study, and met the study criteria. The net participant count to be included in the sample will be determined within the current selection criteria and after the G Powers analysis. The sample size of the study was determined by the post. doc. The sample size will be clarified. With the simple randomization method, students will be assigned to the experimental and control groups. Even the last digit of the student number will be randomized to the experimental group and odd ones will be randomized to the control group Sample Selection Criteria In the sample, it will be considered that virtual reality users may be exposed to strong psychological effects. Discomforts that occur in virtual experiences, which are seen as motion sickness or simulation disease, are among these effects. Simulation hospital is similar to transportation sickness but going through VR experience. It is recommended that motion sickness arises from the accumulation of visual and vestibular senses as its organization. It is seen as headache, fatigue, heaviness, and disorientation in the weight given with the common perception. Advances in Head-Weared Device (HMD) technology may have increased motion sickness enclosures due to increased consumers and levels of realism in virtual reality.

Independent variables

1. Mataverse-based clinical skills lab
2. Socio-demographic characteristics of the people within the scope of the research (age, place of residence, education level of parents)
3. Health status related to technological variables related to people
4. Presence in experimental or control environments
5. Professional development
6. The nature of learning
7. Resources used Designing the Software The software designed by the developers within the Unreal Engine program will first be tested by experts and necessary corrections will be made. The software will be developed in accordance with the design-based research method steps. This method is a research method established to design and develop an evidence-based educational intervention (for example, learning processes, learning environments, etc.) as a solution to an educational problem (teaching-learning strategies and materials, products) (van den Akker et al., 2013). In the design, the student will be presented with the training of a premature baby feeding on a virtual screen with an empty platform, then he will enter the hospital room, evaluate the feeding pattern of the baby in the case and practice appropriate clinical skills.

Expert Evaluation Expert opinion will be taken for the efficiency, suitability, validity, and reliability of the metaverse-based clinical skills laboratory used in the study. Experts; consist of field experts and engineering experts.

ELIGIBILITY:
Inclusion Criteria:

* Participants who gave written and verbal consent to enter the study
* Students taking and continuing the Child Health and Diseases Nursing course

Exclusion Criteria:

1. Participants who received the 1. Child Health and Diseases nursing training for the 2nd time
2. Participants who did not receive the Child Health and Diseases nursing training
3. Participants with motion sickness
4. Participants with vertigo
5. Participants with middle ear balance problems
6. Participants with Meniere's syndrome
7. Participants with a fear of heights
8. Participants with stomach ailments
9. Participants with eye diseases
10. Participants with other problems
11. Participants withdrawing from the study
12. Participants who dropped out of the study

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-test | one week
  It is a knowledge test that aims to measure the relevant knowledge of the dependent variable before the application and experiment

SECONDARY OUTCOMES:
Final Test | one month
  It is a knowledge test that aims to measure the relevant knowledge of the dependent variable after application and experimentation.
Proficiency Scale for Nursing Students | one month
  By Bektaş, Bektaş, and Ayar (2020) Pediatric Nursing Proficiency Scale for Nursing Students: After reviewing existing research and receiving relevant faculty input, researchers created it for nursing students to evaluate pediatric nursing competencies.
Augmented Reality Applications Attitude Scale | one month
  "Augmented Reality Attitude Scale" The scale, which was developed by Küçük, Yılmaz, Baydaş, and Göktaş (2014) and whose validity and reliability was made, consists of 15 items in a 5-point Likert scale.
Focus Group Interview Form | one month
  A focus group interview is a qualitative data collection method, which is generally held with 4-12 participants and a moderator and aims to collect data by creating a polyphonic environment where participants do not need to hide their true thoughts.
Distance Education Satisfaction Scale of university life | one month
  "University Students' Distance Education Satisfaction Scale" The scale, which was developed by Kafes and Yıldırım (2021), and whose validity and reliability was established, consists of 8 items in a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Kuğuoğlu, Prof. Dr., Study Chair — Medipol University

IPD SHARING:
Plan to Share IPD: No